CLINICAL TRIAL: NCT04419090
Title: Cascade Genetic Testing of Familial Hypercholesterolemia: the CATCH Multicenter Randomized Controlled Trial
Brief Title: Cascade Genetic Testing of Familial Hypercholesterolemia
Acronym: CATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Swiss Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020-01271
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Monogenic positive FH, direct contact (Experimental)
  Interventions: Other: web-based centralized service and message
- Monogenic positive FH, usual care (No Intervention)
- Monogenic negative FH, direct contact (Experimental)
  Interventions: Other: web-based centralized service and message
- Monogenic negative FH, usual care (No Intervention)

INTERVENTIONS:
Other: web-based centralized service and message — Perform three cycles of cascade screening through several generation of family members of an index case. The contact of relatives will be initiated by the index case and supported by a web-based centralized service. The index case will be provided with a prepared email or Whatsapp message that the index case can further forward to his first-degree relatives. The email/message will contain a link to a secured web application with a code for the connection. By clicking on the link, the relative will connect to a specifically designed app. The app will provide information about the transmission mode of FH, the cardiovascular risk associated with FH and the way how to reduce this risk. The relative can then fill out information and provide agreement to be contacted for the study. The nearest specialized clinic will then contact the relative to organize further screening with similar processes.
  Arms: Monogenic negative FH, direct contact; Monogenic positive FH, direct contact

SUMMARY:
Familial hypercholesterolemia (FH) is a frequent genetic disorder (1/200) associated with an increased risk of early-onset myocardial infarction. To improve detection and treatment of patient with FH, cascade genetic testing in families is recommended by many cardiovascular prevention guidelines. However, the implementation of national genetic cascade screening is challenging, because legal protection to guarantee privacy of data do not authorize physicians to directly contact at-risk relatives. Using current mobile information technologies and a centralized web-based platform, we designed an ethical genetic cascade screening program for FH to be tested in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe hypercholesterolemia and familial or personal history of early-onset cardiovascular disease = Dutch Lipid Clinic Network score (DLNC) >= 6 points.

Exclusion Criteria:

* Patients without at least one contactable first-degree family members

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
the yield of detection of familial hypercholesterolemia (FH) | 2 years
  The yield of detection is the number of test performed/number of contactable relatives.

CONTACTS AND LOCATIONS:
Overall Officials: David Nanchen, MD, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Locations (1):
- Center for primary care and public health (Unisanté), University of Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided